CLINICAL TRIAL: NCT05609201
Title: PRospective Evaluation of Interstitial Lung DIsease Progression With Quantitative CT
Acronym: PREDICT-ILD
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: North Bristol NHS Trust (Other); Royal United Hospitals Bath NHS Foundation Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-22-54
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each time point the following blood samples will be required:
  1. 5ml EDTA for FBC
  2. 5ml SST for CRP
  3. 10ml EDTA for plasma, buffy coat and red blood cell layers for study of peripheral leucocyte telomere length and ELISA for endothelial glycocalyx and angiogenesis markers
  4. 10ml EDTA and 10ml Plasma for stored sample for future ancillary research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 36 participants with a multidisciplinary team diagnosis of IPF or non-IPF fibrotic-ILD
  Interventions: Diagnostic Test: HRCT Thorax; Device: Glycocheck Endothelial Glycocalyx Assessment; Diagnostic Test: Blood biomarkers; Diagnostic Test: Peripheral leucocyte telomere length; Diagnostic Test: Pulmonary function testing; Diagnostic Test: Patient reported outcome measures
- Healthy Control: 5 Age, sex and ethnicity matched controls
  Interventions: Device: Glycocheck Endothelial Glycocalyx Assessment; Diagnostic Test: Blood biomarkers; Diagnostic Test: Peripheral leucocyte telomere length

INTERVENTIONS:
Diagnostic Test: HRCT Thorax — HRCT Thorax at 0, 6 and 12 months
  Groups: Cases
Device: Glycocheck Endothelial Glycocalyx Assessment — Measure of EG degradation using GlycoCheck Microvascular Health Score at 0, 6 and 12 months
Diagnostic Test: Blood biomarkers — Endothelial glycocalyx degradation blood biomarkers and angiogenesis markers at 0, 6 and 12 months
Diagnostic Test: Peripheral leucocyte telomere length — HT-STELA (High-throughput single telomere length assessment) at 0, 6 and 12 months
Diagnostic Test: Pulmonary function testing — Pulmonary Function Tests (Spirometry and Gas Transfer) and 6-minute walk distance at 0, 6 and 12 months
  Groups: Cases
Diagnostic Test: Patient reported outcome measures — Electronic collection of patient reported outcome measures
  Groups: Cases

SUMMARY:
The interstitial lung diseases (ILD) are a heterogenous group of conditions with varying degrees of inflammation and scarring (fibrosis) of the lungs. ILD progression is unpredictable, making prognostication challenging. A proportion of patients will develop inexorably progressive disease termed progressive fibrosing ILD (PF-ILD).

Forced vital capacity (FVC), a lung function variable, is routinely used to monitor disease progression. However FVC can be a poor disease marker as it can be influenced by patient effort and can be difficult to perform. High resolution computed tomography (HRCT) is a necessary investigation for suspected fibrotic-ILD, making it a promising tool for research.

A quantitative-CT (qCT) approach uses computer software to analyse HRCT scans and has advantage over visual radiologist assessments which are limited by inter/intra-observer variance. The investigators will undertake a feasibility study to determine whether baseline and longitudinal qCT can predict and quantify disease progression in fibrotic-ILD.

The endothelial glycocalyx (EG) is a mesh-like layer that lines the small blood vessels. Injury to this layer has been implicated in non-thoracic fibrotic diseases. Telomeres are repetitive genetic sequences which cap chromosomes preventing their damage during cell replication. Prematurely shortened leucocyte telomere lengths (LTL) have been demonstrated in a wide range of ILDs. We will evaluate role of measuring EG health and LTL in disease prognostication.

Adult participants with fibrotic-ILD from 3 centres in England will be recruited alongside healthy controls. Case (disease) participants will undergo investigations at 0, 6 and 12 months from recruitment including:

* HRCT with quantitative analysis (qCT)
* Lung function testing
* EG and LTL measurement
* Health related quality of life assessments

The primary outcome will assess the correlation of disease progression status measured by standard of care (FVC) with baseline qCT and EG assessment. Healthy controls will only undergo EG assessment at all time points. Feasibility outcomes will be assessed including recruitment, consent and attrition rates.

The results will inform a subsequent multi-centre study to assess the clinical benefit of disease monitoring with the measures assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Multidisciplinary team diagnosis of IPF or non-IPF fibrotic-ILD
* Treatment naivety to anti-fibrotic therapy at entry to study
* Adult ≥18 years <85
* Informed consent

Exclusion Criteria:

* Forced expiratory volume in 1s/FVC <0.7,
* Significant other respiratory pathology including emphysema >15% on CT (radiologist determined)
* Evidence of ILD exacerbation at the time of CT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants under the clinical care of the interstitial lung disease teams at the following hospitals:
  * Royal University Hospitals Bath NHS Foundation Trust, UK
  * Royal Devon University Healthcare, UK
  * North Bristol NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of disease progression using multi-modal assessment | 12 months
  Correlation of disease progression status (progressor vs non-progressor) with baseline markers including:
  1. Endothelial glycocalyx health via GlycoCheckTM and blood biomarkers
  2. qCT metrics
  3. Peripheral leucocyte telomere length measured via HT-STELA
Feasibility of using qCT for disease prognostication and monitoring | 12 months
  Recruitment, consent and attrition rates and dropout reasons
Endothelial glycocalyx | 12 months
  III. Comparison of endothelial glycocalyx health between healthy controls and participants with fibrotic interstitial lung disease

SECONDARY OUTCOMES:
Longitudinal disease progression | 12 months
  Correlation of longitudinal change of pulmonary function testing:
  1. Endothelial glycocalyx health via GlycoCheckTM and blood biomarkers
  2. qCT metrics
  3. Peripheral leucocyte telomere length measured via HT-STELA
Exploratory mechanisms | 12 months
  Exploratory analysis of the data to infer causal mechanisms of disease progression
Prediction of disease progression | 12 months
  III. Exploratory analysis of the ability of 6 month qCT and PFT change to predict progression at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Giles Dixon, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter Medical School, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available on an anonymised basis via Open Research Exeter data depository (https://ore.exeter.ac.uk/repository).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Study protocol will be available at the time of study recruitment Informed consent for will be available at the time of study recruitment. Clinical study report will be published within 12 months of study completion.